CLINICAL TRIAL: NCT05984875
Title: The Immune Landscape of Epithelial Ovarian Cancer: a Prospective Observational Study
Brief Title: The Immune Landscape of Epithelial Ovarian Cancer
Acronym: IOSI-GYNE-001
Status: Recruiting | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Institute of Oncology Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOSI-GYNE-001
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- A: Newly diagnosed high grade serous or endometroid OC undergoing primary debulking surgery
  Interventions: Other: Collection of tumor samples, blood and vaginal and rectal swabs
- B: Newly diagnosed high grade serous or endometroid OC undergoing NACT followed by interval debulking surgery. This cohort also includes patients that will not be deemed suitable for interval debulking surgery following NACT
  Interventions: Other: Collection of tumor samples, blood and vaginal and rectal swabs
- C: Rare subtypes of epithelial OC (low grade serous, low grade endometrioid, clear cell, mucinous or carcinosarcoma) undergoing primary debulking surgery
  Interventions: Other: Collection of tumor samples, blood and vaginal and rectal swabs
- D: Rare subtypes of epithelial OC (low grade serous, low grade endometrioid, clear cell, mucinous or carcinosarcoma) undergoing NACT followed by interval debulking surgery. This cohort also includes patients with the selected histological subtypes that will not be deemed suitable to interval debulking surgery following NACT
  Interventions: Other: Collection of tumor samples, blood and vaginal and rectal swabs
- E: Women undergoing adnexectomy for benign pathology

INTERVENTIONS:
Other: Collection of tumor samples, blood and vaginal and rectal swabs — The following biological samples will be collected at different time points, according to the specified cohort and after signing the inform consent form: tumor tissue (fresh and archival) or normal tissue (cohort E), ascites (when present), peripheral blood, rectal swab, vaginal swab.
  Groups: A; B; C; D

SUMMARY:
This is a single center prospective observational study to characterize the immune landscape of newly diagnosed epithelial ovarian cancer (OC).

Patients with newly diagnosed epithelial OC will be enrolled in 4 different cohorts: A) Newly diagnosed high grade serous or endometroid OC undergoing primary debulking surgery; B) Newly diagnosed high grade serous or endometroid OC undergoing neoadjuvant chemotherapy (NACT) followed by interval debulking surgery; C) Rare subtypes of epithelial OC (low grade serous, low grade endometrioid, clear cell, mucinous or carcinosarcoma) undergoing primary debulking surgery; D) Rare subtypes of epithelial OC (low grade serous, low grade endometrioid, clear cell, mucinous or carcinosarcoma) undergoing NACT followed by interval debulking surgery. A cohort of women undergoing adnexectomy for benign pathology will be enrolled (cohort E) for comparative analysis.

Enrolled patients will be asked to provide the following biological samples at specified time points: archival and fresh tumor tissue, peripheral blood samples, rectal and vaginal swabs, ascites (when present).

The main aim of the study is to characterize the immune landscape of epithelial OC in tumor tissue and peripheral blood and correlate the presence of myeloid-derived suppressive cells (MDSCs) and other immune infiltrates and of the systemic immune response with progression free interval (PFI) in epithelial OC.

ELIGIBILITY:
Inclusion criteria cohort A-D:

* Suspicious diagnosis of epithelial ovarian cancer (subsequent histologically confirmation required)
* Plan to undergo a surgical procedure for the management of epithelial ovarian cancer or recurrent ovarian cancer previously treated with conventional treatment and involved in the trial as group A-D
* ≥18 years old
* ECOG Performance Status ≤ 2
* Written informed consent

Inclusion criteria cohort E:

* Indication for adnexectomy for a benign gynecological condition
* ≥18 years old
* ECOG Performance Status ≤ 2
* Written informed consent

Exclusion criteria cohort A-E:

* Other active concomitant neoplasms that might confound the results of the planned analysis.
* Ongoing active autoimmune disease requiring treatment or condition of immune deficiency
* Ongoing chronic treatment with steroids or other immune suppressive agents at the time of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed epithelial ovarian cancer and subjects with bening gynecological conditions requiring surgery
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of the immune cells infiltrate | At the time of diagnosis in the tumor tissue and on blood. For patients receiving chemotherapy, assessment on blood after cycle 3 and 6
  Expression of multiple immune cell markers will be assessed in samples from different subtypes of epithelial ovarian cancer by flow cytometric analysis. Percentages of individual immune cell populations among total tumor-infiltrating immune cells will be evaluated.

SECONDARY OUTCOMES:
To define the prognostic value of the immune cells infiltrate | From diagnosis until disease progression or study termination, whichever will occur first
  The prognostic value of the immune cell populations identified by flow cytometry will be evaluated by calculating the correlation coefficient between the percentage of the immune cell population and the progression-free interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No